CLINICAL TRIAL: NCT06464718
Title: Effectiveness of Calcium and Vitamin D, With and Without Collagen Peptide, in Enhancing Bone Mineral Density on Postmenopausal Women With Osteopenia: Pilot Randomized Controlled Trial.
Brief Title: Effectiveness of Calcium and Vitamin D, With and Without Collagen Peptide, in Enhancing Bone Mineral Density on Postmenopausal Women With Osteopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frontier Medical and Dental College, Abbotabad (Other)
Responsible Party: Principal Investigator, Dr Saif ur Rehman, Professor, Frontier Medical and Dental College, Abbotabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3390
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Osteopenia
Keywords: Bone mineral density; collagen peptide; osteoporosis; osteopenia; vitamin D3
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Intervention Model Description: Group A comprised of 15 subject who were given daily sachet containing 5g of Bio active collagen peptides (Fortibone). Electrolyte mix containing 500 mg calcium as calcium lactate, 4 MCg calcitriol and selenised yeast rich in vitamin D3 (400IU) (Colabone®, Vivapharm SA). Group B (control) consisted of 15 subjects who consumed a sweet formed from a chewable tablet with 1. A calcium compound containing 25 g calcium carbonate (500mg elemental calcium) and vitamin D3 400IU taken daily, these are potent supplements that are often used in practice, as per the researchers' recommendations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fortibone (Experimental)
  Interventions: Drug: Fortibone
- Chewable Tablet (Active Comparator)
  Interventions: Drug: Chewable Tablet

INTERVENTIONS:
Drug: Fortibone — Participants were given daily sachet containing 5g of Bio active collagen peptides (Fortibone). Electrolyte mix containing 500 mg calcium as calcium lactate, 4 MCg calcitriol and selenised yeast rich in vitamin D3 (400IU) (Colabone®, Vivapharm SA).
  Arms: Fortibone
Drug: Chewable Tablet — calcium compound containing 25 g calcium carbonate (500mg elemental calcium) and vitamin D3 400IU taken daily
  Arms: Chewable Tablet

SUMMARY:
Osteopenia is characterized by bone mineral density (BMD) being lower than normal but not reaching the osteoporosis threshold, poses a serious problem for women after menopause. Osteopenia is a precursor to osteoporosis that is associated with increased risk of fractures, morbidity, and mortality. Using strategies to improve or maintain bone density is important for preventing osteoporosis and its associated complications. The combination of collagen peptide (CP) with calcium and vitamin D supplementation may provide several ways to improve bone health. This study aims to provide preliminary evidence of the effectiveness of traditional medicine in improving bone health through the effectiveness of CP.

DETAILED DESCRIPTION:
Osteopenia is characterized by bone mineral density (BMD) being lower than normal but not reaching the osteoporosis threshold, poses a serious problem for women after menopause. Osteopenia is a precursor to osteoporosis that is associated with increased risk of fractures, morbidity, and mortality. Using strategies to improve or maintain bone density is important for preventing osteoporosis and its associated complications. The combination of collagen peptide (CP) with calcium and vitamin D supplementation may provide several ways to improve bone health. This study aims to provide preliminary evidence of the effectiveness of traditional medicine in improving bone health through the effectiveness of CP.The study was single blinded randomized controlled trial, involving 30 post-menopausal women that were equally divided into two groups by computer generated simple random sampling technique. Group A received bioactive collagen peptide along with calcium lactate, and vitamin D3. The control group (Group B) consisted of 15 participants who were given a chewable tablet daily, containing 1.25 grams of calcium carbonate (equivalent to 500 mg of elemental calcium) and 400 IU of vitamin D3.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal patients
* (-1. 0>T-score>-2. 5)

Exclusion Criteria:

* fracture,
* primary hyperparathyroidism

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal
Enrollment: 30 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Blood Test | baseline and after 3 months
  Calcium levels in blood
Blood Test | baseline and after 3 months
  Vitamin B
Blood Test | baseline and after 3 months
  Osteocalcin
Dexa Scan | baseline and after 3 months
  Bone Mineral Density

CONTACTS AND LOCATIONS:
Locations (1):
- Frontier Medical and Dental College, Abbottābād, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No